CLINICAL TRIAL: NCT01613612
Title: Control Study of Implantation of Enriched Bone Marrow Cells for the Treatment of Avascular Necrosis of Femoral Head
Brief Title: Implantation of Bone Marrow Cells to Treat Avascular Necrosis of Femoral Head (ANFH)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Qiujiang Zheng, Director of Orthopaedic Surgery, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GGH_201112_Ortho_1
Record Dates: First submitted 2011-12-13; First posted 2012-06-07 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Avascular Necrosis of Femur Head
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group:core decompression (Sham Comparator): single core decompression
  Interventions: Procedure: core decompression
- Treatment group: BMCs+core decompression (Active Comparator): Enriched bone marrow cells combined with core decompression
  Interventions: Procedure: Enriched BMCs implantation combined with core decompression

INTERVENTIONS:
Procedure: core decompression — minimal surgical invention to drill a core to the femoral head to release pressure
  Arms: control group:core decompression
Procedure: Enriched BMCs implantation combined with core decompression — Patients are subjected to bone marrow aspiration from the anterior iliac crest. Mononuclear cells are enriched from patients' bone marrow by centrifuge, which are grafted with autologous cortical bone and implanted to the necrotic zone of the femoral head.
  Arms: Treatment group: BMCs+core decompression

SUMMARY:
The purpose of this study is to compare the efficacy of autologous enriched bone marrow cell implantation combined with core decompression to single core decompression for the treatment of avascular necrosis of femoral head.

ELIGIBILITY:
Inclusion Criteria:

* femoral head necrosis patients
* stage I/II/III (Ficat)
* age from 18 to 55 years
* stop steroid treatment for minimal 6 months

Exclusion Criteria:

* age younger than 18 or older than 55
* any hemopathy
* tumor
* femoral head/neck fracture

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
change of Visual Analogue Scale | before invention and 24 months after invention
  Change from baseline in 24 months
change of lequensne algofunctional index | before invention and 24 months after invention
  change from baseline in 24 months
change of WOMAC index | before invention and 24 months after invention
  change from baseline in 24 months

REFERENCES:
- [Derived] Li M, Ma Y, Fu G, Zhang R, Li Q, Deng Z, Zheng M, Zheng Q. 10-year follow-up results of the prospective, double-blinded, randomized, controlled study on autologous bone marrow buffy coat grafting combined with core decompression in patients with avascular necrosis of the femoral head. Stem Cell Res Ther. 2020 Jul 16;11(1):287. doi: 10.1186/s13287-020-01810-8. PMID 32678055
- [Derived] Ma Y, Wang T, Liao J, Gu H, Lin X, Jiang Q, Bulsara MK, Zheng M, Zheng Q. Efficacy of autologous bone marrow buffy coat grafting combined with core decompression in patients with avascular necrosis of femoral head: a prospective, double-blinded, randomized, controlled study. Stem Cell Res Ther. 2014 Oct 14;5(5):115. doi: 10.1186/scrt505. PMID 25315149